CLINICAL TRIAL: NCT04123821
Title: The Routine Use of Nasopharyngeal Airway in the Setting of Monitored Anesthesia Care During Gastrointestinal Endoscopy: A Multi-center Randomized Controlled Trial
Brief Title: The Routine Use of Nasopharyngeal Airway in the Setting of Monitored Anesthesia Care During Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Christian Rouphael, Instructor of Clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2018-0549
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Monitored Anesthesia Care; Gastrointestinal Endoscopy; Nasopharyngeal Airway

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Nasopharyngeal airway with 5L/min oxygen through nasal cannula
  Interventions: Device: Nasopharyngeal airway
- Group B (No Intervention): 5 L/min oxygen through nasal cannula alone

INTERVENTIONS:
Device: Nasopharyngeal airway — A disposable nasopharyngeal airway of appropriate size will be selected for patients allocated to the intervention group with 5L/min oxygen through nasal cannula
  Arms: Group A

SUMMARY:
The goal of this prospective, multi-center, single-blinded randomized controlled trial is to assess the efficacy of NPA in reducing respiratory events in patients being admitted for GI endoscopy (colonoscopy, gastroscopy, endoscopic ultrasound) under deep sedation. The main question it aims to answer are: • [Is the NPA used on patients undergoing gastrointestinal endoscopy efficient in reducing respiratory events?] Participants will be randomly allocated into one of the two groups: NPA with 5L/min oxygen through nasal cannula (group A) or 5 L/min oxygen through nasal cannula alone (group B). Researchers will compare NPA group to nasal cannula group to see if the routine placement of an NPA can reduce the frequency of airway obstruction, hypoxemic events and airway maneuvers (chin lift, oral airway insertion, and mask-bag ventilation) during endoscopic sedation.

DETAILED DESCRIPTION:
Monitored anesthesia care (MAC) is currently the dominant method of endoscopic sedation for approximately one third of all US gastroenterologists. The popularity and success of MAC can be ascribed to many factors including increased patient turnover and improved patient satisfaction. Patients undergoing MAC maintain spontaneous breathing and routinely receive supplemental oxygen. In case of airway obstruction, additional airway adjuncts may be used such as supraglottic airway devices including oropharyngeal airway, nasopharyngeal airway, laryngeal mask, etc. A nasopharyngeal airway (NPA) is a simple device that can be conveniently inserted into the supraglottic airway to secure an open passage. This is a prospective, multi-center, single-blinded randomized controlled trial designed to evaluate the efficacy of the routine use of NPA in preventing airway obstruction during deep sedation. Patients undergoing gastrointestinal endoscopy under monitored anesthesia care using target-controlled infusion of propofol at AUBMC will be randomly and equally apportioned to the NPA (group A) or nasal cannula group (group B). Episodes of desaturation, airway maneuvers, hemodynamic instability, adverse events related to NPA insertion, duration of the procedure, and the anesthetic dose will be recorded. The satisfaction of the anesthesiologist, gastroenterologist, and patient will be scored. The aim of this study is first to assess the efficacy of NPA in reducing respiratory events, and second, to identify the safety of this device as well as patient, gastroenterologist and anesthesiologist satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing GI endoscopy under MAC using TCI of Propofol
* Patients above 18 years old
* Patient able to give consent
* ASA classification: I, II, III

Exclusion criteria:

* Patients with craniofacial abnormalities
* Patients with a history of recent nasal or cranial bone fracture
* Patients with a history of recent nasal or trans-sphenoidal surgery
* Patients with nasal polyposis
* Patients with a history of epistaxis
* Patients with a history of coagulopathy or on anticoagulation therapy (including patients on Aspirin not stopped 7 days prior to presentation)
* Patients with a history of allergy to Xylometazoline or local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Respiratory events (desaturation) | During the procedure
  oxygen saturation (%)
Incidence of Respiratory events (chin lift/jaw thrust) | During the procedure
  Occurrence of the event (chin lift/jaw thrust):yes or no and the number of episodes if yes
Incidence of Respiratory events (mask-bag ventilation) | During the procedure
  Occurrence of the event (mask-bag ventilation):yes or no and the number of episodes if yes

SECONDARY OUTCOMES:
Intubation | During the procedure
  Occurrence of the event (intubation): yes or no and the number of episodes if yes
Interruptions during the case | During the procedure
  Occurrence of the event (Interruptions during the case): yes or no and the number of episodes if yes
Incidence of hypotension | During the procedure
  Occurrence of the event (SBP<90 mmHg): yes or no and the number of episodes if yes
Bradycardia | During the procedure
  Occurrence of the event (HR<50 beats/min): yes or no and the number of episodes if yes
Epistaxis | During the procedure
  Development of epistaxis: yes or no and the number of episodes if yes
Cough | During the procedure
  Development of cough: yes or no and the number of episodes if yes
Laryngospasm | During the procedure
  Development of laryngospasm: yes or no and the number of episodes if yes
Movement impeding procedure | During the procedure
  Patient's movement impeded the procedure :yes or no and the number of episodes if yes
Satisfaction score of the anesthesiologist | Up to 2 hours after the procedure
  Satisfaction score of the anesthesiologist on a numerical rating scale from 0 to 10
Satisfaction score of the proceduralist | Up to 2 hours after the procedure
  Satisfaction score of the proceduralist on a numerical rating scale from 0 to 10
Satisfaction score of the patient | Up to 2 hours after the procedure
  Satisfaction score of the patient on a numerical rating scale from 0 to 10

OTHER OUTCOMES:
Duration of the procedure | During the procedure
  Duration of the procedure in minutes
Total amount of Propofol | During the procedure
  Total amount of Propofol in mg

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rouphael, MD, Principal Investigator — American University of Beirut Medical Center; Rony Al Nawar, MD, Principal Investigator — LAU Medical Center-Rizk Hospital
Locations (1):
- Christian Rouphael, Beirut, Lebanon